CLINICAL TRIAL: NCT05978258
Title: An Observational Study Assessing the Experience of Patients Undergoing Active Cluster Headache Clinical Trials
Brief Title: A Close Examination of Patient Experiences in Cluster Headache Clinical Research
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 81829797
Record Dates: First submitted 2023-07-28; First posted 2023-08-07 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-07

CONDITIONS: Cluster Headache
Keywords: Cluster Headache
MeSH Terms: conditions — Cluster Headache

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Historically, participation in clinical studies is highly skewed towards particular demographic groups of people.

This research will invite several participants to gather a wide range of information on clinical trial experiences for cluster headache patients. The aim of the study is to identify the factors that limit the ability of a person to enroll in, as well as complete a clinical trial for treatment of cluster headache.

The data collected from this study will help improve future outcomes for all cluster headache patients as well as those in under-represented demographic groups.

ELIGIBILITY:
Inclusion Criteria:

* Patient has been diagnosed with cluster headache
* Patient has access to a home internet connection in order to provide regular updates through the course of the study
* Participant must be 18 years of age or older

Exclusion Criteria:

* Patient has an ECOG score of 4 or higher
* Patient is not able to provide consistent digital updates as per study requirements
* Patient does not complete or agree to terms outlined in the Informed Consent Form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cluster headache who are actively considering enrolling in a clinical trial for the said condition, but have not yet completed enrollment and randomization phases.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Rate of patients who decide to enroll in a cluster headache clinical study. | 3 months
Number of cluster headache patients who remain in clinical research until completion. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.
Locations (1):
- Power Life Sciences, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Merli E, Asioli GM, Favoni V, Zenesini C, Mascarella D, Sartori A, Cortelli P, Cevoli S, Pierangeli G. Great occipital nerve long-acting steroid injections in cluster headache therapy: an observational prospective study. J Neurol. 2022 Apr;269(4):2193-2199. doi: 10.1007/s00415-021-10884-0. Epub 2021 Nov 25. PMID 34820736
- [Background] Snoer A, Lund N, Beske R, Hagedorn A, Jensen RH, Barloese M. Cluster headache beyond the pain phase: A prospective study of 500 attacks. Neurology. 2018 Aug 28;91(9):e822-e831. doi: 10.1212/01.wnl.0000542491.92981.03. Epub 2018 Jul 27. PMID 30054443
- [Background] Vigano A, Savastano E, Petolicchio B, Toscano M, De Sanctis R, Maestrini I, Di Piero V. A Study of Clinical Features and Risk Factors of Self-Referring Emergency Department Headache Patients: A Comparison with Headache Center Outpatients. Eur Neurol. 2020;83(1):34-40. doi: 10.1159/000505915. Epub 2020 Mar 10. PMID 32155625

DOCUMENTS (1):
  • Informed Consent Form (2023-07-28): https://cdn.clinicaltrials.gov/large-docs/58/NCT05978258/ICF_000.pdf